CLINICAL TRIAL: NCT07330843
Title: Évaluation et évolution de l'identité Narrative et de Son Lien Avec le Bien-être Multidimensionnel Subjectif et le rétablissement Multidimensionnel Dans le Premier épisode Psychotique
Brief Title: Assessment and Evolution of Narrative Identity and Its Relationship to Subjective Multidimensional Well-being and Multidimensional Recovery in First Episode Psychosis
Acronym: PEPID
Status: Not yet recruiting | Type: Observational
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Other Study IDs: LOCAL/2025/THESE/JJ-01
Record Dates: First submitted 2025-12-18; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Psychosis; Mental Disorder
Keywords: Narrative identity
MeSH Terms: conditions — Psychotic Disorders; Mental Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- First episode psychosis
  Interventions: Other: Narrative identity task
- Chronic: participants diagnosed with a psychotic disorder
  Interventions: Other: Narrative identity task
- Control
  Interventions: Other: Narrative identity task

INTERVENTIONS:
Other: Narrative identity task — Participants will be asked to elaborate five personal narratives in response to the different types of questions: trauma, transgression, negative memory, self-definition, and turning point.

SUMMARY:
First episode psychosis (FEP) constitutes an important subgroup within psychotic disorders, as the acute impact of a disorder at the time of diagnosis may differ from its long-term impact over the following decades. Narrative is identified as a sense of personal agency, of belonging to a social group, metacognition, and well-being. Patients with schizophrenia have lower levels of agency and communion compared to HIV-positive participants. However, the themes of agency and communion and metacognition do not reflect all factors representing narrative identity. In order to measure well-being, it is also necessary to introduce a specific and multidimensional measure that will allow a more precise understanding of the phenomenon.

In FEP, a link has been demonstrated between the specificity of self-recollection and functional outcomes. Given that the transitional developmental stage between adolescence and adulthood is a key developmental window for narrative identity as well as psychotic disorders and that narrative identity is positively associated with mental health, this study will therefore focus on the acquisition of narrative identity in the FEP. It will investigate the extent to which narrative identity has an impact on multidimensional subjective well-being and whether it can predict multidimensional subjective well-being over time. The study investigators hypothesize that the levels of the various components of narrative identity would be lower in cases of FEP compared to patients with other "chronic" psychotic conditions and controls.

ELIGIBILITY:
Inclusion Criteria:

* Subject who has given their free and informed consent.
* Subject who has signed the consent form.
* Subject who is a member of or beneficiary of a health insurance plan.

For the FEP group:

* Patient treated in a psychiatric department (consultation or hospitalization) for a FEP defined by:
* Presence of positive psychotic symptoms (delusions and/or hallucinations and/or conceptual disorganization) evolving for at least one week, either every day or at least 3 times a week for at least one hour per occasion
* Never having taken neuroleptic treatment with an antipsychotic purpose (with the exception of antipsychotic treatment initiated for the current episode)
* Disorder meeting DSM 5 criteria from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific schizophrenia spectrum disorder or other psychotic disorder, bipolar disorder I or II with mood-congruent and mood-incongruent psychotic features, substance-induced bipolar disorder with mood-congruent and mood-incongruent psychotic features, major depressive disorder with mood-congruent and mood-incongruent psychotic features

For the "Chronic" group:

• Patients diagnosed with a disorder meeting DSM-5 criteria for more than 18 months from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophreniform disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific schizophrenia spectrum disorder or other psychotic disorder, bipolar I or II disorder with mood-congruent and mood-incongruent psychotic features, substance-induced bipolar disorder with mood-congruent and mood-incongruent psychotic features, major depressive disorder with mood-congruent and mood-incongruent psychotic features

Exclusion Criteria:

* The subject is participating in category 1 RIPH or a clinical drug trial or clinical investigation study, or is in a period of exclusion determined by a previous study
* The patient is unable to express consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* Pregnant or breastfeeding subject.
* Patient with a history of traumatic brain injury
* Patient with moderate to severe mental retardation (IQ ≤ 55)

For the FEP group:

• FEP related to a drug-induced psychotic disorder or due to another medical condition

For the "Control" group:

* Patient with lifetime experience of FEP
* Patient with a diagnosis of a disorder meeting DSM-5 criteria from the following list: delusional disorder, brief psychotic disorder lasting more than 7 days, schizophrenia-like disorder, schizophrenia, schizoaffective disorder, substance-induced psychotic disorder lasting more than 7 days, other specific or non-specific schizophrenia spectrum disorder or other psychotic disorder, bipolar I or II disorder with mood-congruent and mood-incongruent psychotic features, bipolar disorder with mood-congruent and mood-incongruent psychotic features substance-induced mood, major depressive disorder with psychotic features congruent and incongruent with mood

Ages: 16 Years to 30 Years | Sex: All
Age Groups: Child, Adult
Study Population: 406 / 5,000
  Three groups of participants will be formed:
  1. a group of participants meeting the criteria for a FEP;
  2. a group of "chronic" participants diagnosed with a psychotic disorder (recruited from patients at the Carémeau University Hospital in Nîmes); and
  3. a control group of participants, representative of the general population (recruited through social media advertisements).
Sampling Method: Non-Probability Sample
Enrollment: 96 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2029-07 (Estimated); Study Completion 2029-07 (Estimated)

PRIMARY OUTCOMES:
Emotional valence according to the question: "When you think about this story in your life, how positive or negative is this story in your life?" | Baseline (Day 0)
  7-point scale ranging from -3 "Extremely negative" to 3 "Extremely positive"
Emotional valence according to the question: "When you think about this story in your life, how positive or negative is this story in your life?" | Month 6
  7-point scale ranging from -3 "Extremely negative" to 3 "Extremely positive"
Emotional valence according to the question: "When you think about this story in your life, how positive or negative is this story in your life?" | Month 12
  7-point scale ranging from -3 "Extremely negative" to 3 "Extremely positive"
Emotional valence according to the question: "When you think about this story in your life, how positive or negative is this story in your life?" | Month 18
  7-point scale ranging from -3 "Extremely negative" to 3 "Extremely positive"
Emotional valence according to the question: "When you think about this story in your life, how positive or negative is this story in your life?" | Month 24
  7-point scale ranging from -3 "Extremely negative" to 3 "Extremely positive"
Emotional intensity according to the question: "When you think about this story in your life, how intense is this story in your life?" | Baseline (Day 0)
  7-point scale ranging from 1 "Not at all intense" to 7 "Extremely intense" -
Emotional intensity according to the question: "When you think about this story in your life, how intense is this story in your life?" | Month 6
  7-point scale ranging from 1 "Not at all intense" to 7 "Extremely intense" -
Emotional intensity according to the question: "When you think about this story in your life, how intense is this story in your life?" | Month 12
  7-point scale ranging from 1 "Not at all intense" to 7 "Extremely intense" -
Emotional intensity according to the question: "When you think about this story in your life, how intense is this story in your life?" | Month 18
  7-point scale ranging from 1 "Not at all intense" to 7 "Extremely intense" -
Emotional intensity according to the question: "When you think about this story in your life, how intense is this story in your life?" | Month 24
  7-point scale ranging from 1 "Not at all intense" to 7 "Extremely intense" -
Emotional tone according to the question "When you think about this story in your life, is it generally negative, mixed, neutral, or positive?" | Baseline (day 0)
  4-point scale ranging from 0 "Negative" to 4 "Positive."
Emotional tone according to the question "When you think about this story in your life, is it generally negative, mixed, neutral, or positive?" | Month 6
  4-point scale ranging from 0 "Negative" to 4 "Positive."
Emotional tone according to the question "When you think about this story in your life, is it generally negative, mixed, neutral, or positive?" | Month 12
  4-point scale ranging from 0 "Negative" to 4 "Positive."
Emotional tone according to the question "When you think about this story in your life, is it generally negative, mixed, neutral, or positive?" | Month 18
  4-point scale ranging from 0 "Negative" to 4 "Positive."
Emotional tone according to the question "When you think about this story in your life, is it generally negative, mixed, neutral, or positive?" | Month 24
  4-point scale ranging from 0 "Negative" to 4 "Positive."

SECONDARY OUTCOMES:
Narrative identity between groups | Baseline (Day 0)
  PERMA Profiler questionnaire; a 15-item scale in which higher scores indicate greater well-being
Narrative identity between groups | Month 6
  PERMA Profiler questionnaire; a 15-item scale in which higher scores indicate greater well-being
Narrative identity between groups | Month 12
  PERMA Profiler questionnaire; a 15-item scale in which higher scores indicate greater well-being
Narrative identity between groups | Month 18
  PERMA Profiler questionnaire; a 15-item scale in which higher scores indicate greater well-being
Narrative identity between groups | Month 24
  PERMA Profiler questionnaire; a 15-item scale in which higher scores indicate greater well-being
General health-related quality of life between groups | Baseline (day 0)
  EQ5D-5L questionnaire comprising five items representing the five dimensions, and a visual analog scale ranging from 0 to 100 (100 referring to the "best possible health state"). The responses are then into a 5-digit number describing the patient's health state (e.g "11111" indicates the absence of problems).
General health-related quality of life between groups | Month 6
  EQ5D-5L questionnaire comprising five items representing the five dimensions, and a visual analog scale ranging from 0 to 100 (100 referring to the "best possible health state"). The responses are then into a 5-digit number describing the patient's health state (e.g "11111" indicates the absence of problems).
General health-related quality of life between groups | Month 12
  EQ5D-5L questionnaire comprising five items representing the five dimensions, and a visual analog scale ranging from 0 to 100 (100 referring to the "best possible health state"). The responses are then into a 5-digit number describing the patient's health state (e.g "11111" indicates the absence of problems).
General health-related quality of life between groups | Month 18
  EQ5D-5L questionnaire comprising five items representing the five dimensions, and a visual analog scale ranging from 0 to 100 (100 referring to the "best possible health state"). The responses are then into a 5-digit number describing the patient's health state (e.g "11111" indicates the absence of problems).
General health-related quality of life between groups | Month 24
  EQ5D-5L questionnaire comprising five items representing the five dimensions, and a visual analog scale ranging from 0 to 100 (100 referring to the "best possible health state"). The responses are then into a 5-digit number describing the patient's health state (e.g "11111" indicates the absence of problems).
Health-related quality of life between groups | Baseline (day 0)
  WHOQOL-Brief: a 26-item questionnaire including one item on overall quality of life, one item assessing general health, and one item from each of the 24 facets of the WHOQOL-100. Four types of five-point response scales measure intensity (Not at all-Extremely), capacity (Not at all-Completely), frequency (Never-Always), and evaluation (Very dissatisfied/Very poor-Very satisfied/Very good).
Health-related quality of life between groups | Month 6
  WHOQOL-Brief: a 26-item questionnaire including one item on overall quality of life, one item assessing general health, and one item from each of the 24 facets of the WHOQOL-100. Four types of five-point response scales measure intensity (Not at all-Extremely), capacity (Not at all-Completely), frequency (Never-Always), and evaluation (Very dissatisfied/Very poor-Very satisfied/Very good).
Health-related quality of life between groups | Month 12
  WHOQOL-Brief: a 26-item questionnaire including one item on overall quality of life, one item assessing general health, and one item from each of the 24 facets of the WHOQOL-100. Four types of five-point response scales measure intensity (Not at all-Extremely), capacity (Not at all-Completely), frequency (Never-Always), and evaluation (Very dissatisfied/Very poor-Very satisfied/Very good).
Health-related quality of life between groups | Month 18
  WHOQOL-Brief: a 26-item questionnaire including one item on overall quality of life, one item assessing general health, and one item from each of the 24 facets of the WHOQOL-100. Four types of five-point response scales measure intensity (Not at all-Extremely), capacity (Not at all-Completely), frequency (Never-Always), and evaluation (Very dissatisfied/Very poor-Very satisfied/Very good).
Health-related quality of life between groups | Month 24
  WHOQOL-Brief: a 26-item questionnaire including one item on overall quality of life, one item assessing general health, and one item from each of the 24 facets of the WHOQOL-100. Four types of five-point response scales measure intensity (Not at all-Extremely), capacity (Not at all-Completely), frequency (Never-Always), and evaluation (Very dissatisfied/Very poor-Very satisfied/Very good).
Anxiety and depression between groups | Baseline (Day 0)
  Hospital Anxiety and Depression Scale questionnaire where a higher score indicates greater distress
Anxiety and depression between groups | Month 6
  Hospital Anxiety and Depression Scale questionnaire where a higher score indicates greater distress
Anxiety and depression between groups | Month 12
  Hospital Anxiety and Depression Scale questionnaire where a higher score indicates greater distress
Anxiety and depression between groups | Month 18
  Hospital Anxiety and Depression Scale questionnaire where a higher score indicates greater distress
Anxiety and depression between groups | Month 24
  Hospital Anxiety and Depression Scale questionnaire where a higher score indicates greater distress
Autobiographical memory between groups | Baseline (day 0)
  Thinking About Life Experiences scale (TALE-15): 17-item questionnaire consists of two general questions followed by 15 specific items related to the functions of autobiographical memory, each composed of 5 sub-items. Responses are rated on a 5-point Likert scale ranging from "Almost never" to "Very frequently."
Autobiographical memory between groups | Month 6
  Thinking About Life Experiences scale (TALE-15): 17-item questionnaire consists of two general questions followed by 15 specific items related to the functions of autobiographical memory, each composed of 5 sub-items. Responses are rated on a 5-point Likert scale ranging from "Almost never" to "Very frequently."
Autobiographical memory between groups | Month 12
  Thinking About Life Experiences scale (TALE-15): 17-item questionnaire consists of two general questions followed by 15 specific items related to the functions of autobiographical memory, each composed of 5 sub-items. Responses are rated on a 5-point Likert scale ranging from "Almost never" to "Very frequently."
Autobiographical memory between groups | Month 18
  Thinking About Life Experiences scale (TALE-15): 17-item questionnaire consists of two general questions followed by 15 specific items related to the functions of autobiographical memory, each composed of 5 sub-items. Responses are rated on a 5-point Likert scale ranging from "Almost never" to "Very frequently."
Autobiographical memory between groups | Month 24
  Thinking About Life Experiences scale (TALE-15): 17-item questionnaire consists of two general questions followed by 15 specific items related to the functions of autobiographical memory, each composed of 5 sub-items. Responses are rated on a 5-point Likert scale ranging from "Almost never" to "Very frequently."
Personality type between groups | Baseline (day 0)
  Big Five Inventory (BFI-10): assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability, and openness.
Personality type between groups | Month 6
  Big Five Inventory (BFI-10): assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability, and openness.
Personality type between groups | Month 12
  Big Five Inventory (BFI-10): assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability, and openness.
Personality type between groups | Month 18
  Big Five Inventory (BFI-10): assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability, and openness.
Personality type between groups | Month 24
  Big Five Inventory (BFI-10): assessing the five major personality traits: extraversion, agreeableness, conscientiousness, emotional stability, and openness.
Symptomatology of psychotic disorders in the FEP and chronic groups | Baseline (day 0)
  Positive and negative symptom scale (PANSS). 30 items measuring 5 subscales: positive, negative, disorganization, hostility, and anxiety. Each item is rated on a 7-point Likert scale ranging from 1 (absent) to 7 (extreme). The positive subscale ranges from 7 to 49, the negative subscale from 8 to 56, the hostility subscale from 6 to 46, the disorganization subscale from 5 to 35, and the anxiety subscale from 4 to 28. The total score ranges from 30 to 210.
Symptomatology of psychotic disorders in the FEP and chronic groups | Month 6
  Positive and negative symptom scale (PANSS). 30 items measuring 5 subscales: positive, negative, disorganization, hostility, and anxiety. Each item is rated on a 7-point Likert scale ranging from 1 (absent) to 7 (extreme). The positive subscale ranges from 7 to 49, the negative subscale from 8 to 56, the hostility subscale from 6 to 46, the disorganization subscale from 5 to 35, and the anxiety subscale from 4 to 28. The total score ranges from 30 to 210.
Symptomatology of psychotic disorders in the FEP and chronic groups | Month 12
  Positive and negative symptom scale (PANSS). 30 items measuring 5 subscales: positive, negative, disorganization, hostility, and anxiety. Each item is rated on a 7-point Likert scale ranging from 1 (absent) to 7 (extreme). The positive subscale ranges from 7 to 49, the negative subscale from 8 to 56, the hostility subscale from 6 to 46, the disorganization subscale from 5 to 35, and the anxiety subscale from 4 to 28. The total score ranges from 30 to 210.
Symptomatology of psychotic disorders in the FEP and chronic groups | Month 18
  Positive and negative symptom scale (PANSS). 30 items measuring 5 subscales: positive, negative, disorganization, hostility, and anxiety. Each item is rated on a 7-point Likert scale ranging from 1 (absent) to 7 (extreme). The positive subscale ranges from 7 to 49, the negative subscale from 8 to 56, the hostility subscale from 6 to 46, the disorganization subscale from 5 to 35, and the anxiety subscale from 4 to 28. The total score ranges from 30 to 210.
Symptomatology of psychotic disorders in the FEP and chronic groups | Month 24
  Positive and negative symptom scale (PANSS). 30 items measuring 5 subscales: positive, negative, disorganization, hostility, and anxiety. Each item is rated on a 7-point Likert scale ranging from 1 (absent) to 7 (extreme). The positive subscale ranges from 7 to 49, the negative subscale from 8 to 56, the hostility subscale from 6 to 46, the disorganization subscale from 5 to 35, and the anxiety subscale from 4 to 28. The total score ranges from 30 to 210.
Overall functioning in the FEP and chronic groups | Baseline (day 0)
  Global Assessment of Functioning (GAF). This numerical scale (from 0 to 100) subjectively assesses functioning in social, occupational, and psychological domains. Lower scores represent lower levels of functioning
Overall functioning in the FEP and chronic groups | Month 6
  Global Assessment of Functioning (GAF). This numerical scale (from 0 to 100) subjectively assesses functioning in social, occupational, and psychological domains. Lower scores represent lower levels of functioning
Overall functioning in the FEP and chronic groups | Month 12
  Global Assessment of Functioning (GAF). This numerical scale (from 0 to 100) subjectively assesses functioning in social, occupational, and psychological domains. Lower scores represent lower levels of functioning
Overall functioning in the FEP and chronic groups | Month 18
  Global Assessment of Functioning (GAF). This numerical scale (from 0 to 100) subjectively assesses functioning in social, occupational, and psychological domains. Lower scores represent lower levels of functioning
Overall functioning in the FEP and chronic groups | Month 24
  Global Assessment of Functioning (GAF). This numerical scale (from 0 to 100) subjectively assesses functioning in social, occupational, and psychological domains. Lower scores represent lower levels of functioning
Personal recovery in the FEP and chronic groups | Baseline (day 0)
  Stage of recovery instrument (STORI): a 50-item questionnaire that evaluates the five stages of personal recovery. Ten themes are assessed, each containing five items ranging from 0 "Not at all true" to 5 "Completely true," corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50
Personal recovery in the FEP and chronic groups | Month 6
  Stage of recovery instrument (STORI): a 50-item questionnaire that evaluates the five stages of personal recovery. Ten themes are assessed, each containing five items ranging from 0 "Not at all true" to 5 "Completely true," corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50
Personal recovery in the FEP and chronic groups | Month 12
  Stage of recovery instrument (STORI): a 50-item questionnaire that evaluates the five stages of personal recovery. Ten themes are assessed, each containing five items ranging from 0 "Not at all true" to 5 "Completely true," corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50
Personal recovery in the FEP and chronic groups | Month 18
  Stage of recovery instrument (STORI): a 50-item questionnaire that evaluates the five stages of personal recovery. Ten themes are assessed, each containing five items ranging from 0 "Not at all true" to 5 "Completely true," corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50
Personal recovery in the FEP and chronic groups | Month 24
  Stage of recovery instrument (STORI): a 50-item questionnaire that evaluates the five stages of personal recovery. Ten themes are assessed, each containing five items ranging from 0 "Not at all true" to 5 "Completely true," corresponding to the five stages of personal recovery. A score is calculated for each stage, ranging from 0 to 50
Social and individual performance in the FEP and chronic groups | Baseline (day 0)
  Personal and social performance scale (PSP): measures four domains of social and individual functioning (socially useful activities, personal and social relationships, self-care, disruptive and aggressive behaviors) and provides a score between 1 and 100, divided into 10 equal intervals to assess the degree of difficulty. Higher scores correspond to better personal and social functioning, with scores of 91 to 100 indicating more than adequate functioning, while scores below 30 indicate such poor functioning that intensive supervision is required.
Social and individual performance in the FEP and chronic groups | Month 6
  Personal and social performance scale (PSP): measures four domains of social and individual functioning (socially useful activities, personal and social relationships, self-care, disruptive and aggressive behaviors) and provides a score between 1 and 100, divided into 10 equal intervals to assess the degree of difficulty. Higher scores correspond to better personal and social functioning, with scores of 91 to 100 indicating more than adequate functioning, while scores below 30 indicate such poor functioning that intensive supervision is required.
Social and individual performance in the FEP and chronic groups | Month 12
  Personal and social performance scale (PSP): measures four domains of social and individual functioning (socially useful activities, personal and social relationships, self-care, disruptive and aggressive behaviors) and provides a score between 1 and 100, divided into 10 equal intervals to assess the degree of difficulty. Higher scores correspond to better personal and social functioning, with scores of 91 to 100 indicating more than adequate functioning, while scores below 30 indicate such poor functioning that intensive supervision is required.
Social and individual performance in the FEP and chronic groups | Month 18
  Personal and social performance scale (PSP): measures four domains of social and individual functioning (socially useful activities, personal and social relationships, self-care, disruptive and aggressive behaviors) and provides a score between 1 and 100, divided into 10 equal intervals to assess the degree of difficulty. Higher scores correspond to better personal and social functioning, with scores of 91 to 100 indicating more than adequate functioning, while scores below 30 indicate such poor functioning that intensive supervision is required.
Social and individual performance in the FEP and chronic groups | Month 24
  Personal and social performance scale (PSP): measures four domains of social and individual functioning (socially useful activities, personal and social relationships, self-care, disruptive and aggressive behaviors) and provides a score between 1 and 100, divided into 10 equal intervals to assess the degree of difficulty. Higher scores correspond to better personal and social functioning, with scores of 91 to 100 indicating more than adequate functioning, while scores below 30 indicate such poor functioning that intensive supervision is required.
Improvement of clinical state in the FEP and chronic groups | Baseline (day 0)
  Clinical global impression (CGI): a global observer-rated assessment tool that measures a patient's clinical condition before and after medical treatment. It consists of two measures: Severity, which measures the severity of the patient's clinical condition; and Improvement, which assesses the improvement in the patient's clinical condition since the start of treatment, both on a scale of 1 to 7.
Improvement of clinical state in the FEP and chronic groups | Month 6
  Clinical global impression (CGI): a global observer-rated assessment tool that measures a patient's clinical condition before and after medical treatment. It consists of two measures: Severity, which measures the severity of the patient's clinical condition; and Improvement, which assesses the improvement in the patient's clinical condition since the start of treatment, both on a scale of 1 to 7.
Improvement of clinical state in the FEP and chronic groups | Month 12
  Clinical global impression (CGI): a global observer-rated assessment tool that measures a patient's clinical condition before and after medical treatment. It consists of two measures: Severity, which measures the severity of the patient's clinical condition; and Improvement, which assesses the improvement in the patient's clinical condition since the start of treatment, both on a scale of 1 to 7.
Improvement of clinical state in the FEP and chronic groups | Month 18
  Clinical global impression (CGI): a global observer-rated assessment tool that measures a patient's clinical condition before and after medical treatment. It consists of two measures: Severity, which measures the severity of the patient's clinical condition; and Improvement, which assesses the improvement in the patient's clinical condition since the start of treatment, both on a scale of 1 to 7.
Improvement of clinical state in the FEP and chronic groups | Month 24
  Clinical global impression (CGI): a global observer-rated assessment tool that measures a patient's clinical condition before and after medical treatment. It consists of two measures: Severity, which measures the severity of the patient's clinical condition; and Improvement, which assesses the improvement in the patient's clinical condition since the start of treatment, both on a scale of 1 to 7.
Awareness of the disorders in the FEP and chronic groups | Baseline (day 0)
  Birchwood insight scale (BIS); multidimensional assessment of awareness of illness (insight) and includes 8 questions (3-point Likert scale: "agree," "disagree," or "uncertain"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Awareness of the disorders in the FEP and chronic groups | Month 6
  Birchwood insight scale (BIS); multidimensional assessment of awareness of illness (insight) and includes 8 questions (3-point Likert scale: "agree," "disagree," or "uncertain"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Awareness of the disorders in the FEP and chronic groups | Month 12
  Birchwood insight scale (BIS); multidimensional assessment of awareness of illness (insight) and includes 8 questions (3-point Likert scale: "agree," "disagree," or "uncertain"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Awareness of the disorders in the FEP and chronic groups | Month 18
  Birchwood insight scale (BIS); multidimensional assessment of awareness of illness (insight) and includes 8 questions (3-point Likert scale: "agree," "disagree," or "uncertain"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Awareness of the disorders in the FEP and chronic groups | Month 24
  Birchwood insight scale (BIS); multidimensional assessment of awareness of illness (insight) and includes 8 questions (3-point Likert scale: "agree," "disagree," or "uncertain"). The overall score ranges from 0 to 12, with a score above 9 indicating good insight.
Abstract verbal reasoning in the FEP and chronic groups | Baseline (day 0)
  Similarities section of the Wechsler Adult Intelligence Scale (WAIS): For 18 pairs of words, the participant subject must identify the qualitative relationship between the two words
Abstract verbal reasoning in the FEP and chronic groups | Month 6
  Similarities section of the Wechsler Adult Intelligence Scale (WAIS): For 18 pairs of words, the participant subject must identify the qualitative relationship between the two words
Abstract verbal reasoning in the FEP and chronic groups | Month 12
  Similarities section of the Wechsler Adult Intelligence Scale (WAIS): For 18 pairs of words, the participant subject must identify the qualitative relationship between the two words
Abstract verbal reasoning in the FEP and chronic groups | Month 18
  Similarities section of the Wechsler Adult Intelligence Scale (WAIS): For 18 pairs of words, the participant subject must identify the qualitative relationship between the two words
Abstract verbal reasoning in the FEP and chronic groups | Month 24
  Similarities section of the Wechsler Adult Intelligence Scale (WAIS): For 18 pairs of words, the participant subject must identify the qualitative relationship between the two words
Non-verbal abstract problem solving in the FEP and chronic groups | Baseline (day 0)
  Matrix reasoning section of the Wechsler Adult Intelligence Scale (WAIS); in which participants must identify patterns in drawings
Non-verbal abstract problem solving in the FEP and chronic groups | Month 6
  Matrix reasoning section of the Wechsler Adult Intelligence Scale (WAIS); in which participants must identify patterns in drawings
Non-verbal abstract problem solving in the FEP and chronic groups | Month 12
  Matrix reasoning section of the Wechsler Adult Intelligence Scale (WAIS); in which participants must identify patterns in drawings
Non-verbal abstract problem solving in the FEP and chronic groups | Month 18
  Matrix reasoning section of the Wechsler Adult Intelligence Scale (WAIS); in which participants must identify patterns in drawings
Non-verbal abstract problem solving in the FEP and chronic groups | Month 24
  Matrix reasoning section of the Wechsler Adult Intelligence Scale (WAIS); in which participants must identify patterns in drawings
Treatment adherence in the FEP and chronic groups | Baseline (day 0)
  Medication adherence rating scale (MARS): 10-item questionnaire concerning medication adherence during the past week assessing behaviors, attitudes, and experiences related to the treatment.
Treatment adherence in the FEP and chronic groups | Month 6
  Medication adherence rating scale (MARS): 10-item questionnaire concerning medication adherence during the past week assessing behaviors, attitudes, and experiences related to the treatment.
Treatment adherence in the FEP and chronic groups | Month 12
  Medication adherence rating scale (MARS): 10-item questionnaire concerning medication adherence during the past week assessing behaviors, attitudes, and experiences related to the treatment.
Treatment adherence in the FEP and chronic groups | Month 18
  Medication adherence rating scale (MARS): 10-item questionnaire concerning medication adherence during the past week assessing behaviors, attitudes, and experiences related to the treatment.
Treatment adherence in the FEP and chronic groups | Month 24
  Medication adherence rating scale (MARS): 10-item questionnaire concerning medication adherence during the past week assessing behaviors, attitudes, and experiences related to the treatment.
Episodic memory between groups | Baseline (day 0)
  California Verbal Learning Test--Second Edition (CVLT): in this word list recall and recognition test, the examiner reads a list of 16 nouns aloud at one-second intervals in a fixed order over five learning trials. The participant is asked to recall as many words as possible in any order (free recall). If subjects "cluster" words from each category, they are presumably using semantic organization. Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall).
Episodic memory between groups | Month 6
  California Verbal Learning Test--Second Edition (CVLT): in this word list recall and recognition test, the examiner reads a list of 16 nouns aloud at one-second intervals in a fixed order over five learning trials. The participant is asked to recall as many words as possible in any order (free recall). If subjects "cluster" words from each category, they are presumably using semantic organization. Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall).
Episodic memory between groups | Month 12
  California Verbal Learning Test--Second Edition (CVLT): in this word list recall and recognition test, the examiner reads a list of 16 nouns aloud at one-second intervals in a fixed order over five learning trials. The participant is asked to recall as many words as possible in any order (free recall). If subjects "cluster" words from each category, they are presumably using semantic organization. Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall).
Episodic memory between groups | Month 18
  California Verbal Learning Test--Second Edition (CVLT): in this word list recall and recognition test, the examiner reads a list of 16 nouns aloud at one-second intervals in a fixed order over five learning trials. The participant is asked to recall as many words as possible in any order (free recall). If subjects "cluster" words from each category, they are presumably using semantic organization. Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall).
Episodic memory between groups | Month 24
  California Verbal Learning Test--Second Edition (CVLT): in this word list recall and recognition test, the examiner reads a list of 16 nouns aloud at one-second intervals in a fixed order over five learning trials. The participant is asked to recall as many words as possible in any order (free recall). If subjects "cluster" words from each category, they are presumably using semantic organization. Free recall is tested immediately (short-term recall) and again after 20 minutes (long-term recall).

CONTACTS AND LOCATIONS:
Overall Officials: Julie Jourdan, Principal Investigator — Centre Hospitalier Universitaire de Nīmes
Locations (1):
- CHU de Nîmes, Nîmes, France